CLINICAL TRIAL: NCT02264730
Title: Phase 1 Single-Arm Study Evaluating ClotFoam as an Adjunct to Hemostasis in Abdominal Surgery in Which Liver Bleeding is Encountered
Brief Title: ClotFoam as an Adjunct to Hemostasis in Abdominal Surgery - Liver Bleeding is Encountered
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biomedica Management Corporation (Industry)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, George Falus, President, Biomedica Management Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-030H2
Record Dates: First submitted 2014-10-06; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clot Foam (Experimental): Application of Clotfoam
  Interventions: Drug: ClotFoam

INTERVENTIONS:
Drug: ClotFoam — Patient has not received blood products between screenings
  Other Names: No other names

SUMMARY:
Phase 1 Single-Arm Study Evaluating ClotFoam as an Adjunct to Hemostasis in Abdominal Surgery in Which Liver Bleeding is Encountered.

DETAILED DESCRIPTION:
In any open surgery bleeding usually occurs. Surgeons try to stop the bleeding by using his/her usual surgical practice. These include, but are not limited to: suturing (stitches), ligation (tying up) or cautery (to burn in order to stop or prevent bleeding). It is often necessary for surgeons to use an additional treatment to stop the bleeding. This may include the use of a hemostatic product (used to stop bleeding).

This Phase I study consists of a single arm evaluating the safety of ClotFoam as an adjunct to hemostasis. ClotFoam® is an investigational product-a gelatin-based hydrogel carrying a fibrin monomer-that has been designed for supportive treatment in general surgery for the improvement of hemostasis, where standard techniques are insufficient.

The evaluation will be conducted in 24 patients who are scheduled to undergo elective open surgery in which liver bleeding is encountered requiring control of mild-to- moderate bleeding where standard surgical techniques are expected to be ineffective and/or impractical. All subjects who meet eligibility criteria and who provide informed consent to participate will be assigned to ClotFoam topical treatment. Subjects who will be screened for eligibility to participate in this study will be those who are scheduled to with undergo an elective (non-emergency) hepatic wedge resection or anatomic resection (of 1 to 5 contiguous hepatic segments or a surgical procedure in which liver bleeding is encountered such as removal of the gall bladder (open), bile duct excision wherein an appropriate target bleeding site is identified.

Subjects undergoing living-related liver donation are also eligible. Participants will have post-operative follow ups at day 1,2,5, and 10 post-procedure, 2 weeks post procedure, and 12 weeks post-procedure. The follow up visits will consist of safety evaluations (physical exam, adverse event assessment, laboratory evaluations).

ELIGIBILITY:
Inclusion Criteria:

* Subject is expected to survive 6 months from the date of screening, If female and of child-bearing potential, subject has a negative serum pregnancy test prior to surgery and agrees to not breast feed her child (if applicable) for duration of study treatment and completion of study follow-up visits, If subject is a sexually active male or a sexually active female of child-bearing potential, subject agrees to use a medically accepted form of contraception from the time of consent to completion of all follow-up study visits

Exclusion Criteria:

* pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
control mild-to-moderate bleeding during surgery in which liver bleeding in encountered | 12 weeks
  evaluated intermittently during those 12 weeks

SECONDARY OUTCOMES:
Hemostatic Success | 1 minute
  Percentage of subjects who achieve hemostatic success within the 1-minute TTH assessment period.
Hemostatic Success | 5 minutes
  Percentage of subjects who achieve hemostatic success within the 5-minute TTH assessment period.
Hemostatic Success | 10 minutes
  Percentage of subjects who achieve hemostatic success within the 10- minute TTH period.
Hemostatic Success | 10 minutes
  Incidence of treatment failures (if hemostasis is not achieved within 10 minutes or if bleeding required additional intervention during the 2nd 10 minute observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Grant Bochicchio, MD, MPH FACS, Principal Investigator — Washington University School of Medicine Barnes Jewish Hospital
Locations (1):
- Washington University School of Medicine Barnes Jewish Hospital Clinical Laboratory, St Louis, Missouri, United States

REFERENCES:
- [Derived] Maegele M. Effective approaches to address noncompressible torso hemorrhage. Curr Opin Crit Care. 2024 Jun 1;30(3):202-208. doi: 10.1097/MCC.0000000000001141. Epub 2024 Feb 28. PMID 38441108